CLINICAL TRIAL: NCT00367718
Title: A Phase II Trial of VELCADE in Patients With Metastatic or Locally Recurrent Nasopharyngeal Carcinoma
Brief Title: Trial of VELCADE in Patients With Metastatic or Locally Recurrent Nasopharyngeal Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left JHU and is not able to be reached for updates
Sponsor: Johns Hopkins University (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRG-NP04/23/06
Record Dates: First submitted 2006-08-21; First posted 2006-08-23 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2019-05

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Bortezomib

INTERVENTIONS:
Drug: Velcade — velcade 1.3 mg/m2 given at the day 1,4,8,and 11 every 21 days schedule.

SUMMARY:
This study seeks to test the Efficacy in terms of rates of disease response in metastatic nasopharyngeal carcinoma of the standard dose of velcade 1.3 mg/m2 given at the day 1,4,8,and 11 every 21 days schedule. The study uses a Simons 2 stage design and will enroll between 15-25 patients. Secondary endpoints studied include Pharmacokinetics, toxicities, EBV viral load and molecular characterization of EBV in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven nasopharyngeal carcinoma - WHO type 3 (recurrence or metastases)
* metastatic disease or locally recurrent disease not amendable curative therapy
* Patients must have measurable disease
* least one (not more than a total of three prior lines of chemotherapy for metastatic or recurrent disease). This must include at least 1 prior line of platinum-containing chemotherapy.
* An ECOG performance status of 0-2
* Absolute neutrophil count (ANC) ≥1500/mm3
* Hemoglobin 8g/dl (blood transfusion is allowed to correct hemoglobin level).
* PLT ≥ 75,000/mm 3
* Total bilirubin ≤ 2 x upper normal limit (UNL)
* Serum ALT ≤ 5 x UNL
* Serum creatinine ≤ 2 mg/dL
* Serum albumin ≥ 2.5 g/dL
* No known history of brain or leptomeningeal metastasis.
* ≥ 18 years of age.
* Estimated life expectancy ≥ 24 weeks.
* For sexually active women of childbearing potential, negative pregnancy test within 21 days of enrolling on trial.
* must be able to give informed written consent

Exclusion Criteria:

* Patients who have not had at least 1 or more than 3 previous lines of treatment for metastatic or recurrent NPC
* Prior BORTEZOMIB therapy
* Immunotherapy ≤ 4 weeks have elapsed prior to study entry
* Biologic therapy ≤ 4 weeks have elapsed prior to study entry
* Radiation therapy ≤ 4 weeks have elapsed prior to study entry
* Major surgery, or significant traumatic injury ≤3 weeks prior to study entry
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any other therapy or supportive care considered investigational
* Evidence of CNS involvement
* Presence of > grade 1 sensory peripheral neuropathy of any etiology OR grade 1 with neuropathic pain of any etiology.
* Patients with significant local symptoms from metastases which is amenable to radiotherapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BORTEZOMIB.
* History of other malignancy ≤ 3 years prior to study entry, except for adequately treated basal cell, squamous cell skin cancer or cervical intraepithelial neoplasia.
* Uncontrolled intercurrent illness
* Patients who are pregnant or breast feeding (Sexually active men and women of childbearing potential must use contraception during course of therapy and within 3 months of completion of trial) Participation in another clinical trial involving therapeutic intervention within 4 weeks of enrollment.
* Known history of HIV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Efficacy based on response of measurable disease | duration of study (4 -6 months)

SECONDARY OUTCOMES:
EBV viral load | duration of study (4 -6 months)
toxicities | duration of study (4 -6 months)
molecular characterization of EBV in Plasma | duration of study (4 -6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-son Hsieh, M.D., Study Chair — Johns Hopkins Singapore-International Medical Center; Brigette Ma, M.D., Study Chair — Chinese University of Hong Kong
Locations (3):
- Chinese University of Hong Kong, Hong Kong, China
- Singapore (2):
  - Johns Hopkin Singapore International Medical Center, Singapore
  - National University Hospital of Singapore, Singapore